CLINICAL TRIAL: NCT00499044
Title: CDR Versus MATRICS Cognitive Batteries in Patients With Schizophrenia
Brief Title: A Comparison of Two Cognitive Batteries in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Responsible Party: A. Eden Evins, M.D., M.P.H., Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CORRC #18-2007
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: cognition; attention; memory; concentration; schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MATRICS Consensus Cognitive Battery
  Interventions: Other: MATRICS Consensus Cognitive Battery
- 2 (Experimental): Cognitive Drug Research Computerized Cognitive Assessment System
  Interventions: Other: CDR Computerized Cognitive Assessment System

INTERVENTIONS:
Other: CDR Computerized Cognitive Assessment System — Cognitive Drug Research Computerized Cognitive Assessment System consists of performance tasks that measure reaction time, numeric and spatial working memory, word and picture recall and recognition, and episodic secondary memory. CDR is a single, unified battery that can be stored and administered using a laptop computer.
  Other Names: CDR
  Arms: 2
Other: MATRICS Consensus Cognitive Battery — The MATRICS Consensus Cognitive Battery measures functioning across various cognitive domains, such as attention, working memory (verbal and nonverbal), learning (verbal and visual), reasoning and problem solving, and social cognition. Its measurements are based on timed paper-and-pencil, computerized, and orally-administered tests, as well as spatial tests using geometric cubes.
  Other Names: MCCB; MATRICS
  Arms: 1

SUMMARY:
The investigators will compare the test-retest reliabilities of two cognitive batteries in people with schizophrenia: Cognitive Drug Research Computerized Cognitive Assessment System ("CDR") and MATRICS Consensus Cognitive Battery ("MCCB"). The investigators hypothesize that there will be a statistically significant difference in the test-retest reliabilities between MCCB and CDR. In addition, the investigators hypothesize that each of the two batteries will better measure certain areas of cognition. The investigators also hypothesize that scores from both batteries will correlate with quality of life scores, and that there will be a significant difference between the correlations of MCCB and CDR. The investigators hypothesize there will be a significant difference in patients' self-reported tolerability and satisfaction of the MATRICS versus CDR assessments. Lastly, the investigators hypothesize that there will be a significant difference in the MATRICS versus CDR batteries with respect to an administrator-rated score of practicality.

Approximately 32 subjects will enroll in the study. Following consent and eligibility screening (visit 1) and baseline clinical assessment and training in the use of the CDR battery (visit 2), subjects will be randomized into one of two groups for visits 3 and 4. One group will complete the CDR and then MCCB in visit 3, as well as the Tolerability Scale for each battery. The other group will complete the batteries in reverse order during visit 3. Each group will complete both batteries again in reverse order for visit 4. Randomization will be done in blocks of 2. After completion of every 4 subjects, study administrators will complete the Practicality Scale for each battery.

DETAILED DESCRIPTION:
The National Institute of Mental Health's Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) program was a collaboration between members of academia, industry, and the government, with the goal of furthering the development of drugs for the treatment of the cognitive deficits of schizophrenia. The program led to the creation of the MATRICS Consensus Cognitive Battery (MCCB), which measures functioning across various cognitive domains, such as attention, working memory (verbal and nonverbal), learning (verbal and visual), reasoning and problem solving, and social cognition. Its measurements are based on timed paper and pencil, computerized, and orally administered tests, as well as spatial tests using geometric cubes.

Cognitive Drug Research (CDR) is a United Kingdom-based company that has developed another battery of assessments capable of measuring cognitive function in patients with schizophrenia. Its Computerized Cognitive Assessment System consists of performance tasks that measure reaction time, numeric and spatial working memory, word and picture recall and recognition, and episodic secondary memory. CDR is a single, unified battery that can be stored and administered using a laptop computer.

Cognitive assessments are important in establishing the efficacy of medications and other therapeutic interventions for improving cognitive function in patients with schizophrenia. Furthermore, this cognitive functioning is correlated with patients' ability to operate in the real world. This study aims to examine the test-retest reliabilities of the CDR and MATRICS cognitive batteries, and thereby gauge their value for use in studies of cognitive functioning in people with schizophrenia. The investigators hypothesize that for patients with schizophrenia there will be a significant difference in the test-retest reliabilities between the two batteries. Additional aims are to investigate the extent to which MCCB and CDR measure functioning in specific cognitive domains and to investigate patient tolerability and overall practicality of each battery.

Visit 1 (1.5 hours): Baseline Measures and Screening

* Consent
* Review of medical chart to confirm DSM-IV diagnosis of schizophrenia/schizoaffective disorder (depressed type) and medical/psychiatric stability
* Demographic questionnaire
* Salivary drug test to exclude current use of PCP, cannabis, alcohol, cocaine, amphetamine, methamphetamine, and opiates

Visit 2 (2 hours): Clinical Assessment and Training

* Clinical Rating Scales: Scale for the Assessment of Negative Symptoms (SANS), Brief Psychiatric Rating Scale (BPRS), Quality of Life Scale (QLS)
* CDR training

Visits 3 and 4 (2.5 hours each): Patients are randomized into one of two groups:

Group 1

* Visit 3: CDR battery followed by MATRICS battery (with short break in between); Tolerability Scale after each battery.
* Visit 4 (two weeks after Visit 3): MATRICS battery followed by CDR battery (with short break in between); Tolerability Scale after each battery.

Group 2

* Visit 3: MATRICS battery followed by CDR battery (with short break in between); Tolerability Scale after each battery.
* Visit 4 (two weeks after Visit 3): CDR battery followed by MATRICS battery (with short break in between); Tolerability Scale after each battery.

Subjects will undergo a screening visit and chart review to assure the clinical appropriateness and safety of their participation. Subjects are free to withdraw from the study at any stage without giving a reason.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged 18-65 with DSM-IV diagnosis of schizophrenia or schizoaffective disorder (depressed type) by diagnostic interview and chart review.
2. Clinically stable on a stable dose of antipsychotic medication for at least one month; no current active suicidal ideation.
3. Not treated with investigational medication in the past 30 days.
4. Competent to provide informed consent.

Exclusion Criteria:

1. Diagnosis of dementia, neurodegenerative disease, seizure disorder, current substance abuse or dependence disorders, including alcohol, active within the last 3 months or any Axis I DSM-IV diagnosis other than schizophrenia or schizoaffective disorder (depressed type).
2. Serious illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease that is not stabilized such that hospitalization for treatment of that illness is likely within the next two months.
3. Patients who, in the investigator's opinion, pose a current severe homicide or suicide risk.
4. History of multiple head injuries with neurological sequelae or a single severe head injury with lasting neurological sequelae.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Test-retest reliabilities of MATRICS Consensus Cognitive Battery (MCCB) and the Cognitive Drug Research (CDR) Computerized Cognitive Assessment System | 4 weeks

SECONDARY OUTCOMES:
Cognitive domains measured by MCCB versus CDR | 4 weeks
Correlation of MCCB versus CDR scores with clinical measures of quality of life | 4 weeks
Self-reported tolerability and satisfaction of the MCCB and CDR assessments | 4 weeks
Practicality of MCCB versus CDR as reported by test administrators | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, M.D., M.P.H., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Freedom Trail Clinic, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Green MF, Kern RS, Heaton RK. Longitudinal studies of cognition and functional outcome in schizophrenia: implications for MATRICS. Schizophr Res. 2004 Dec 15;72(1):41-51. doi: 10.1016/j.schres.2004.09.009. PMID 15531406
- [Background] Andreasen NC. The Scale for the Assessment of Negative Symptoms (SANS): conceptual and theoretical foundations. Br J Psychiatry Suppl. 1989 Nov;(7):49-58. No abstract available. PMID 2695141
- [Background] Heinrichs DW, Hanlon TE, Carpenter WT Jr. The Quality of Life Scale: an instrument for rating the schizophrenic deficit syndrome. Schizophr Bull. 1984;10(3):388-98. doi: 10.1093/schbul/10.3.388. PMID 6474101
- [Background] Cornblatt BA, Risch NJ, Faris G, Friedman D, Erlenmeyer-Kimling L. The Continuous Performance Test, identical pairs version (CPT-IP): I. New findings about sustained attention in normal families. Psychiatry Res. 1988 Nov;26(2):223-38. doi: 10.1016/0165-1781(88)90076-5. PMID 3237915